CLINICAL TRIAL: NCT06171087
Title: Influence of Domperidon on the Experience of Emotions, Brain and Bodily Activity
Brief Title: Emotions, Dopamine, Brain and Body
Acronym: EMBODY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Prof. Dr., German Institute of Human Nutrition
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: Domperidone emotions
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Emotions
MeSH Terms: interventions — Domperidone

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled intervention with 20mg of Domperidon
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Domperidon (Active Comparator): Participants recieve 10mg of Domperidon, 45 minutes before the start of the experiment
  Interventions: Drug: Domperidon
- Placebo (Placebo Comparator): Participants recieve a placebo pill, 45 minutes before the start of the experiment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Domperidon — oral
  Arms: Domperidon
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
The study will examine the influence of domperidon (20mg) on brain and hebavioral responses to emotional stimuli (videos) using fMRI

ELIGIBILITY:
Inclusion criteria

* 18-40 years old men and women
* Consent to participate
* Fluent in German
* Physically and mentally healthy. No regular medication
* BMI 18-25 kg/m2
* Alcohol consumption less than 15 glasses a week (wine / beer, a glass of higher-percentage alcohol counts as two glasses of beer)
* No illegal drug consumption in the week previous to the experiment
* No smoking
* No extreme athletes
* No vegetarians or vegans or any other dietary restrictions due to allergies or intolerances
* Normal day-night rhythm (no shift work)

Exclusion criteria

* Former or current illnesses of:
* Brain or mind (including anxiety disorders, depression, eating disorders, personality disorders, alcohol, drugs or drug dependence, neurological disorders other than occasional headache, psychiatric or neurological abnormalities)
* Heart or blood circulation
* Gastro-intestinal or endocrine disorders
* Other serious past or present medical conditions (for example, metabolic syndrome, diabetes).
* Current medication and medication over a period of two weeks prior to the examination.
* Other serious health problems or present strong mental or physical stress.
* No current infection or excessive stress
* Missing consent to receive information about incidental findings from the MRI
* Tendency to claustrophobia, dizziness or panic attacks.
* Wear a non-removable pacemaker, defibrillator, hearing aid, drug pump, neurostimulator or implant with solenoid valve (e.g., artificial bowel outlet).
* Metal parts or implants inside the body, for example, due to surgery or injury with a metallic foreign object (e.g., hip replacements, artificial joints, heart valves, vessel occlusions or dilatations, surgical clips, bone screws or plates, coil, shunts, catheters, electrodes, coils, radiation sources, shrapnel, projectiles, stents).
* Have non-removable metal parts or metal-containing devices on or in the body.
* Have ferromagnetic metal parts or implants inside the body (e.g., hip replacements, artificial joints, heart valves, vessel occlusions or dilatations, surgical clips, bone screws or plates, coils, shunts, catheters, electrodes, coils, radiation sources, shrapnel, projectiles, stents)
* Wearing magnetically fixed implants (e.g., amalgam fillings, glass eye).
* Professionally or privately being involved in the processing of metals.
* Have large tattoos (whole limbs).
* Being pregnant.
* Wear a intra-uterine device.
* Having tinnitus.
* Hypersensitivity or allergy to Domperidone or common excipients (lactose-1, corn Starch, potato starch, microcrystalline cellulose, castor oil, povidone, sodium lauryl sulfate, magnesium stearate, hypromellose)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Brain responses to emotions | 1-3 hour after drug administratrion
  fMRI brain responses to emotional videos comparing placebo vs domperidon condition. Specifically: dampened brain response to disgust and high arousing videos in domperidon condition
Body (stomach, heart, skin conductance) response to emotions | 1-3 hour after drug administratrion
  Physiological responses to emotional videos comparing placebo vs domperidon condition. Specifically: Reduction in Tachyhastria for disgust and high arousing videos in domperidone condition
Behavioral responses to emotions | 1-3 hour after drug administratrion
  Changes in subjective reports to emotional videos comparing placebo vs domperidon condition. Specifically: Reduction in disgust and arousal ratings to disgust and high arousing videos

CONTACTS AND LOCATIONS:
Locations (1):
- German Institute of Human Nutrition, Potsdam, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided